## Improving Delirium Screening and Detection for Older Adults Presenting to the Emergency Department (ED): A Novel ED Delirium Screening and Detection Program

Information Sheet for Nurse Champions

Principle Investigator: Liron Sinvani, MD NCT05606328 Document Date: 10/28/2022

## **Northwell Health**

## Consent for Participation in a Research Study

**Study Title:** Improving Delirium Screening and Detection for Older Adults Presenting to the Emergency Department (ED): A Novel ED Delirium Screening and Detection Program

**Sponsor:** National Institutes of Health (NIH)

Principal Investigator: Liron Sinvani, MD

## **Research Study Summary:**

- The purpose of this research is to study the potential of an Emergency Department Delirium Detection Program (ED-DDP) to address the need for consistent and accurate ED delirium detection. We will determine the preliminary efficacy of the ED-DDP to improve ED delirium screening, detection, and management for older adults and also evaluate outcomes of the ED-DDP for site staff.
- As a Delirium Champion, you will be asked to participate in a one-day Delirium Champion Training Workshop, 3 tele-training sessions with a member of the study team to receive observation and feedback regarding bedside delirium screening and screening training, and, along with your site's other Delirium Champions, provide bedside delirium screening trainings to the rest of the ED nurses at your site. You will be asked to submit logs for these nurse training sessions so we can track the trainings completed at your site. Your involvement will require approximately 15 hours over the course of 3 months. Study involvement is intended to occur during your scheduled work hours.
- You will not be paid for volunteering to participate as a Delirium Champion in this study.
- The main risk to you in this research is loss of confidentiality. To help us protect your privacy, this research is covered by a Certificate of Confidentiality from the US Department of Health and Human Services. Study information will be stored in a Northwell-approved database to store PHI and only accessible to research staff listed on the approved protocol.
- Study records that may identify you will be kept private. Investigators will share information collected from this research with the study sponsor (National Institutes of Health) and/or its agents, other researchers, accrediting agencies, and our safety officer. Representatives from Federal and state government oversight agencies such as the Department of Health and Human Services and the National Institutes of Health, and representatives from Northwell Health's Human Research Protection Program may inspect and copy records pertaining to this research.
- The study may have no direct benefit to you, however your contributions in this study will inform a larger-scale version of this study in the future. The larger study will examine the impact of the ED-DDP on patient outcomes and will inform a comprehensive program to improve delirium management and outcomes in the emergency department.
- The alternative is not to participate as a Delirium Champion. Taking part in this study is voluntary. You can choose to take part, decline, or change your mind at any time. Your employment and/or standing will not be impacted if you decide not to participate. If you are a patient of Northwell, the quality of your medical care or future care at Northwell Health will not be affected, regardless of your decision, and you will not be penalized or lose benefits to which you are entitled.

Version Date: 10/07/2022 IRB Number: 22-0681

Northwell Health

HRPP APPROVED October 28, 2022

- Information collected from you for this research may be used or shared with other investigators for future research. If this happens, information which could identify you will be removed. Since identifying information will be removed, there will not be an additional consent for future research. By participating in this study, you are agreeing to allow your data to be used by future researchers without additional consent.
- If you have any questions about the study or would like to withdraw, you may call the Clinical Research Coordinator, Alexandra Perrin, at (646) 864-6020.

Version Date: 10/07/2022 IRB Number: 22-0681

